CLINICAL TRIAL: NCT00148967
Title: Inhibition of Unnecessary RV Pacing With AV Search Hysteresis in ICDs
Brief Title: INTRINSIC RV - Inhibition of Unnecessary RV Pacing With AV Search Hysteresis in ICDs
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CR-CA-051403-T
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Last update posted 2006-11-22 (Estimated); Status verified 2006-11

CONDITIONS: Tachycardia
Keywords: right ventricular pacing; implantable cardioverter defibrillator
MeSH Terms: conditions — Tachycardia | interventions — Defibrillators, Implantable

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator

SUMMARY:
INTRINSIC RV is a two-armed randomized trial that will compare the effects of innovative dual-chamber pacing with AV Search Hysteresis to standard VVI among ICD patients.

DETAILED DESCRIPTION:
The purpose of study is to assess whether AVSH will provide benefits of a dual-chamber ICD without the deleterious effects of unnecessary RV pacing. This study will aim to demonstrate that DDDR-AVSH is equal to VVI with respect to mortality and HF hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet VITALITY™AVT® ICD indications
* Patients who sign and date a Patient Informed Consent prior to device implant
* Patients who remain in the clinical care of the enrolling physician

Exclusion Criteria:

* Patients with current indication for CRT-D
* Patients who previously had a pacemaker, ICD or CRT-D
* Patients with chronic AF
* Patients whose life expectancy is <12 months due to other medical conditions
* Patients who are expected to receive a heart transplant during the duration of the study
* Patients with epicardial pacing leads
* Patients who have CABG, PCI, cardiac or other arrhythmia surgery planned but not yet performed
* Patients with or who are likely to receive a tricuspid or other valve prosthesis
* Patients who are currently enrolled in another investigational study that would directly impact the treatment or outcome of the current study
* Patients who are younger than 18 years of age
* Patients who are pregnant
* Patients who are mentally incompetent and cannot give Patient Informed Consent or participate in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 1535
Dates: Start 2003-07; Study Completion 2005-10

PRIMARY OUTCOMES:
Demonstrate that DDDR-AVSH is as effective as VVI with respect to the composite endpoint of death or heart failure hospitalizations.

SECONDARY OUTCOMES:
The following variables will be compared between patients who are randomized to either DDDR-AVSH or VVI:
The prevalence of atrial fibrillation, Changes in medication dosage, including beta-blocker, anti-arrhythmic and coumadin medications, Programming changes, Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Brian Olshansky, MD, Principal Investigator — University of Iowa; John Day, MD, Principal Investigator — Utah Heart Clinic

REFERENCES:
- [Derived] Sullivan RM, Russo AM, Berg KC, Stolen KQ, Seth M, Perschbacher D, Day JD, Olshansky B. Arrhythmia rate distribution and tachyarrhythmia therapy in an ICD population: results from the INTRINSIC RV trial. Heart Rhythm. 2012 Mar;9(3):351-8. doi: 10.1016/j.hrthm.2011.10.018. Epub 2011 Oct 19. PMID 22016074
- [Derived] Ahmadi-Kashani M, Kessler DJ, Day J, Bunch TJ, Stolen KQ, Brown S, Sbaity S, Olshansky B; INTRINSIC RV Study Investigators. Heart rate predicts outcomes in an implantable cardioverter-defibrillator population. Circulation. 2009 Nov 24;120(21):2040-5. doi: 10.1161/CIRCULATIONAHA.108.847608. Epub 2009 Nov 9. PMID 19901194
- [Derived] Bunch TJ, Day JD, Olshansky B, Stolen KQ, Mullin CM; INTRINSIC RV Study Investigators. Newly detected atrial fibrillation in patients with an implantable cardioverter-defibrillator is a strong risk marker of increased mortality. Heart Rhythm. 2009 Jan;6(1):2-8. doi: 10.1016/j.hrthm.2008.09.025. Epub 2008 Sep 27. PMID 18996055